CLINICAL TRIAL: NCT03307382
Title: Evaluation of the Utility of Single-operator Digital Cholangioscopy During Endoscopic Retrograde Cholangiopancreatography in the Diagnosis of Malignant and Benign Biliary Strictures
Brief Title: Single-operator Digital Cholangioscopy for the Diagnosis of Malignant and Benign Biliary Strictures
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond Shing Yan Tang, Clinical Professional Consultant, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SOC for biliary strictrure
Record Dates: First submitted 2017-10-02; First posted 2017-10-11 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Biliary Stricture
Keywords: Biliary stricture, cholangioscopy

STUDY DESIGN:
Intervention Model Description: Cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- SpyGlass DS Cholangioscopy (Experimental): ERCP with cholangiogram will be performed to assess the common bile duct (CBD) and intrahepatic ducts (IHD) for presence of a stricture. Once a biliary stricture is confirmed on cholangiogram during ERCP, SpyGlass DS Cholangioscopy would be performed. The visual impression (VI) of the biliary stricture will be assessed. Tissue acquisition of the biliary stricture will be performed by cholangioscopy directed biopsy (CDBx), and conventional brush cytology with or without intraductal biopsy. Endoscopic stenting will be performed in standard fashion for biliary drainage to relieve the obstructive jaundice.
  Interventions: Device: SpyGlass DS Cholangioscopy

INTERVENTIONS:
Device: SpyGlass DS Cholangioscopy — SpyGlass DS Cholangioscopy includes a 10 French diameter single use digital cholangioscope and a light source with the digital sensor. During ERCP with cholangioscopic exam, the cholangioscope would be first inserted through the working channel of the duodenoscope and subsequently passed into the bile duct for direct visualization of the bile duct mucosa. The visual impression (VI) of the biliary stricture will be assessed. Tissue acquisition of the biliary stricture will be performed by cholangioscopy directed biopsy (CDBx), and conventional brush cytology with or without intraductal biopsy.

SUMMARY:
Differentiation between malignant and benign biliary strictures can be challenging. Accurate differentiation of malignant biliary strictures from benign ones is crucial to guide management decisions.

While conventional tissue acquisition techniques such as brush cytology or intraductal biopsy of the biliary stricture is often performed during ERCP for tissue diagnosis, their sensitivities are suboptimal. The average sensitivities for brush cytology and intraductal biopsy were reported to be ~ 59% and ~ 63% respectively.

When the cause of a biliary stricture remains unclear despite conventional ERCP techniques for diagnosis, cholangioscopy is often performed during ERCP to clarify the diagnosis. This allows an endoscopist to obtain a visual impression (VI) and to perform targeted biopsy under direct visualization of the biliary stricture.

Recently, a digital SOC system (SpyGlass Digital System (SpyGlass DS), Boston Scientific, USA) has become available and has the potential to further improve the diagnosis of malignant and benign biliary strictures. The utility of this digital SOC in the evaluation of biliary strictures has not been well studied. We propose this study to evaluate the utility of the digital SOC during ERCP in the diagnosis of malignant and benign biliary strictures.

DETAILED DESCRIPTION:
Differentiation between malignant and benign biliary strictures can be challenging. Accurate differentiation of malignant biliary strictures from benign ones is crucial to guide management decisions. While a mass lesion involving the bile duct may be observed on imaging such as ultrasound (USG), computed tomography (CT), or magnetic resonance imaging (MRI) in patient presenting with obstructive jaundice, early malignancy of the bile duct may often present with a ductal stricture without an obvious mass on imaging. Diagnosis of early stage malignancy of the bile duct is desirable since the lesion may be amenable to surgical resection of curative intent.

Endoscopic retrograde cholangiopancreatography (ERCP) is an important diagnostic and therapeutic endoscopic technique in patients with obstructive jaundice and a suspected biliary stricture. While conventional tissue acquisition techniques such as brush cytology or intraductal biopsy of the biliary stricture is often performed during ERCP for tissue diagnosis, their sensitivities are suboptimal. The average sensitivities for brush cytology and intraductal biopsy were reported to be ~ 59% and ~ 63% respectively.

When the cause of a biliary stricture remains unclear despite conventional ERCP techniques for diagnosis, cholangioscopy is often performed during ERCP to clarify the diagnosis. Cholangioscopy performed during ERCP involves passing a small scope (~ 10 French in size) through the working channel of the ERCP duodenoscope for direct visualization of the bile duct mucosa. This allows an endoscopist to obtain a visual impression (VI) and to perform targeted biopsy under direct visualization of the biliary stricture. The VI of a malignant biliary stricture is often characterized by the presence of intraductal abnormal tissue growth, and dilated, irregular, tortuous tumor vessels. During standard ERCP, cholangioscopy can be performed using a 2-operator "mother-baby" system, or a single-operator system. While the 2-operator "mother-baby" cholangioscopy technique can provide good image quality of the biliary stricture during ERCP, its use has been limited due to the cumbersome nature of the procedure requiring 2 endoscopists and the relative fragility of the video cholangioscope. Single-operator cholangioscopy (SOC) system, such as the SpyGlass Direct Visualization System, on the other hand allows a single operator to perform cholangioscopy during ERCP. In a recent meta-analysis of the studies using the optical fiber based SOC in the evaluation of indeterminate biliary strictures, the combined sensitivity and specificity of VI were 90% and 87% respectively, and the combined sensitivity and specificity of cholangioscopy directed biopsy were 69% and 98% respectively. The overall incidence of procedure-related adverse event (eg, infection, perforation, pancreatitis, etc) was reported to be 7.5% for diagnostic SOC during ERCP.

Despite the promising results of VI using the optical fiber based SOC from prior studies, the actual image quality in daily clinical practice is frequently regarded as fair only due to the use of a small optical fiber for imaging, and gradual loss of resolution over time from optical fiber damage. A SOC with better image quality is needed for better endoscopic diagnosis of a biliary stricture.

Recently, a digital SOC system (SpyGlass Digital System (SpyGlass DS), Boston Scientific, USA) has become available and has the potential to further improve the diagnosis of malignant and benign biliary strictures. The utility of this digital SOC in the evaluation of biliary strictures has not been well studied. We propose this study to evaluate the utility of the digital SOC during ERCP in the diagnosis of malignant and benign biliary strictures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients presenting with obstructive jaundice with clinical suspicion for a biliary stricture based on imaging findings or during ERCP
* Written informed consent available

Exclusion Criteria:

* Contraindications for endoscopy due to comorbidities
* Unable to provide written informed consent
* Patients with clinical evidence of ongoing cholangitis precluding a safe cholangioscopy procedure
* Pregnant patients
* Moribund patients from terminal illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
sensitivity, specificity, and accuracy of the digital SOC during ERCP in the diagnosis of malignant and benign biliary strictures. | Till a diagnosis of a malignant stricture is made, or follow up period of at least 6 months for presumed benign stricture
  To assess the sensitivity, specificity, and accuracy of digital SOC in the diagnosis of biliary strictures

CONTACTS AND LOCATIONS:
Overall Officials: Raymond S Tang, MD, Principal Investigator — Prince of Wales Hospital, The Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No